CLINICAL TRIAL: NCT02088476
Title: Candidemia in a Pediatric Center and Importance of Central Venous Catheter Removal
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Eda Karadag Oncel, MD, Hacettepe University Department of Pediatric Infectious Diseases, Hacettepe University
Other Study IDs: HUTF06
Record Dates: First submitted 2014-03-10; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Candidemia
Keywords: candidemia; children; mortality; risk factors
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Candidemia: Candidemia is defined as the presence of growth of any candida species in at least one blood culture obtained by either peripheral venipuncture or through an indwelling central venous catheter.

SUMMARY:
Candidemia has emerged as an important cause of hospital-associated blood-stream infection in children. The purpose of this study was to identify differences in distribution of candida species, risk factors, treatment, and clinical outcome of candidemia in children. This study in children ≤18 years with blood culture proven candidemia identified between 2004 and 2012. Analyses included the determination of causative candida species, resistance to antifungals and clinical outcome, as well as the identification of potential risk factors associated with candidemia.

ELIGIBILITY:
Inclusion Criteria:

* Presence of growth of any candida species in at least one blood culture

Exclusion Criteria:

* Febrile neutropenic patients who were using empirical antifungal agents

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with candidemia were included in our hospital between Jan 2004 and Dec 2012.
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2004-01; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Risk factors of candidemia | up to 3 months
  The presence or absence of potential risk factors for candidemia such as an indwelling central venous catheter (CVC), use of antibiotics (administered for >72 hours), use of antifungals (administered for >24 hours), immunosuppressants, total parenteral nutrition (TPN), admission to the intensive care unit (ICU), mechanical ventilation, neutropenia, hypoalbuminemia and hypophosphatemia.

SECONDARY OUTCOMES:
Prognosis according to candida species | up to 3 months
  Death which ensues within 30 days of the onset of candidemia with no apparent alternative cause is recognized as a candidemia-attributable mortality. Patients who died and survived were compared according to candida species (C.albicans, C. parapsilosis, C. tropicalis, C. sake, C.glabrata).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Karadag-Oncel E, Kara A, Ozsurekci Y, Arikan-Akdagli S, Cengiz AB, Ceyhan M, Gur D, Celik M, Ozkaya-Parlakay A. Candidaemia in a paediatric centre and importance of central venous catheter removal. Mycoses. 2015 Mar;58(3):140-8. doi: 10.1111/myc.12288. Epub 2015 Feb 10. PMID 25678411